CLINICAL TRIAL: NCT01423422
Title: Effects of Low Frequency Electromagnetic Field on Patients With Exercise Induced Angina
Brief Title: Effects of Low Frequency Magnetic Field on Exercise Induced Angina
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aerotel Ltd (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: frequency medicine for angina
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Angina Exacerbation Acute
Keywords: Exercise stress test; Effort Angina; Exercise induced angina
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Frequency exposed patients: Patients exposed to the magnetic field with the specific frequency

SUMMARY:
The investigators have previously shown that a frequency of 15.95-16.00 Hz protects against acute myocardial infarction in rats. In the current study the investigators would like to investigate whether this frequency enables cardiac patients with exercise-induced chest pain to exercise at higher workload and heart rate. Therefore, patients will undergo two exercise stress tests, one test after being exposed to 30 minutes of the above mentioned frequency and another test after being exposed to sham (no frequency is turned ON). The investigators will measure changes in the electrocardiogram (ECG), workload, exercise time, and subjective measure of chest pain (angina).

DETAILED DESCRIPTION:
Several studies have shown that low frequency electromagnetic field has biological and therapeutic potential on the human body, however, to very limited extent on the heart. In the current study cardiac patients suffering from exercise-induced-angina will undergo two consecutive stress tests, one test after being exposed for 30 minutes to the magnetic field and the other test after being exposed to placebo (magnetic field not operated). The order of which the magnet will be operated will be randomly assigned for the patients so a group of patients will be exposed to the magnetic field at their first stress test and another groups of patients will be exposed to the magnetic field at their second stress test. During resting period, and while the patients are subjected to the magnetic field, a 12 lead electrocardiogram (ECG) will be monitored. Thereafter the magnetic field and frequency will be turned off and the patients will be subjected to graded exercise stress test during which they will be monitored for ECG and blood pressure changes. Similar monitoring will be documented during the recovery period following the stress test. In addition, the patients will grade their angina score as documented during the stress test. The data will be compared between the two stress tests and to document any advantageous of the magnetic field on exercise time, workload, ECG changes and/or chest pain.

ELIGIBILITY:
Inclusion Criteria:

Patients with known exercise-induced-angina

Exclusion Criteria:

Patients that changed treatment course between the two exercise stress tests Patients that decided to drop from the second exercise stress test

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled at the Cardiac Rehabilitation Institute, sheba Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-05 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Exercise workload for a given ECG change | within a month from the second exercise stress test
  Exercise workload wil be compared between the two tests and according with the ECG changes recorded at these two tests.

SECONDARY OUTCOMES:
Angina scale | Within a month from the last exercise stress test
  Define the angina scale obtained between the two tests at a given workload.

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Hai, MD, Principal Investigator — Cardiac Rehabilitation Institute, Sheba Medical Center
Locations (1):
- Cardiac Rehabilitation Institute, sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Barzelai S, Dayan A, Feinberg MS, Holbova R, Laniado S, Scheinowitz M. Electromagnetic field at 15.95-16 Hz is cardio protective following acute myocardial infarction. Ann Biomed Eng. 2009 Oct;37(10):2093-104. doi: 10.1007/s10439-009-9758-2. Epub 2009 Jul 9. PMID 19588249